CLINICAL TRIAL: NCT00005603
Title: ALinC 17: Protocol for Patients With Newly Diagnosed High Risk Acute Lymphoblastic Leukemia (ALL) - Evaluation of the Augmented BFM Regimen: A Phase III Study
Brief Title: Combination Chemotherapy in Treating Children With Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: 9906; COG-P9906 (Other: Children's Oncology Group); POG-9906 (Other: Pediatric Oncology Group); CDR0000067722 (Other: ClinicalTrials.gov)
Record Dates: First submitted 2000-05-02; First posted 2003-01-27 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Leukemia
Keywords: childhood acute lymphoblastic leukemia in remission; B-cell childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia | interventions — Asparaginase; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Doxorubicin; Mercaptopurine; Methotrexate; Prednisone; Thioguanine; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: asparaginase
Drug: cyclophosphamide
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: dexamethasone
Drug: doxorubicin hydrochloride
Drug: mercaptopurine
Drug: methotrexate
Drug: prednisone
Drug: thioguanine
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one chemotherapy drug may kill more cancer cells. It is not yet known which combination chemotherapy regimen is more effective for acute lymphoblastic leukemia.

PURPOSE: Phase III trial to determine the effectiveness of combination chemotherapy in treating children who have newly diagnosed acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether augmented BFM therapy is superior to ALinc 14/15 therapy in patients with newly diagnosed high-risk acute lymphoblastic leukemia.
* Determine whether minimal residual disease after induction therapy is predictive of an inferior prognosis in this patient population.
* Determine the correlation between event-free survival, minimal residual disease, and early response in this patient population treated with this multiple drug regimen.

OUTLINE: Patients are stratified by CNS or testicular disease (yes vs no).

* Induction therapy (weeks 1-5): Patients receive oral prednisone 3 times daily on days 1-29; vincristine IV on days 1, 8, 15, and 22; daunorubicin IV on days 8, 15, 22; and asparaginase intramuscularly (IM) on days 2, 5, 8, 12, 15, and 19. Patients also receive methotrexate intrathecally (IT) on days 1 and 8. Patients with CNS 2 or 3 disease also receive methotrexate IT on days 15 and 22.

Patients with M1 bone marrow proceed to consolidation therapy. Patients achieving M2 bone marrow on day 29 receive oral prednisone 3 times daily on days 29-42; vincristine IV and daunorubicin IV over 15 minutes on days 29 and 36; and asparaginase IM on days 29, 32, 36, and 39. If bone marrow is M3 on day 29 or M2 on day 43, then patient is off study.

* Consolidation therapy (weeks 6-14): Patients receive cyclophosphamide IV over 30 minutes on days 1 and 29; cytarabine subcutaneously (SC) or IV on days 2-5, 9-12, 30-33, and 37-40; oral mercaptopurine daily on days 1-14 and 29-42; vincristine IV on days 15, 22, 43, and 50; asparaginase IM on days 15, 17, 19, 22, 24, 26, 43, 45, 47, 50, 52, and 54; and methotrexate IT on days 1, 15, 29, and 43.

Patients then proceed to interim maintenance and delayed intensification on weeks 15-46. Courses repeat every 16 weeks.

* Maintenance I and II (weeks 15-22 and 31-38): Patients receive vincristine IV and methotrexate IV on days 1, 11, 21, 31, and 41; asparaginase IM on days 2, 12, 22, 32, and 42; and methotrexate IT on days 1 and 31.
* Delayed Intensification (weeks 23-36 and 39-42): Patients receive vincristine IV on days 57, 64, and 71; methotrexate IT on day 57; oral dexamethasone 2-3 times daily on days 57-63 and 71-77; doxorubicin IV over 15 minutes 3 times weekly on days 57, 64, and 71; and asparaginase IM on days 60, 62, 64, 67, 69, and 71.
* Delayed Intensification-Reconsolidation (weeks 27-30 and 43-46): Patients receive oral thioguanine on days 85-98; methotrexate IT on day 85; cyclophosphamide IV over 30 minutes on day 85; cytarabine IV or SC on days 86-89 and 93-96; asparaginase IM on days 99, 101, 103, 106, 108, and 110; and vincristine IV on days 99 and 106.
* Continuation therapy (weeks 47-130): Patients receive vincristine IV on days 1, 29, and 57; oral dexamethasone twice daily for 5 consecutive days on days 1-5, 29-33, and 57-61; oral mercaptopurine on days 1-84; oral methotrexate on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78; and methotrexate IT on day 1.

Patients with CNS 3 disease or who are within 24 months of diagnosis with an initial WBC ≥ 100,000/mm^3 undergo whole brain radiotherapy (omit or discontinue mercaptopurine and IT methotrexate) on day 1. Testicular radiotherapy also begins on day 1.

Patients may receive oral methotrexate on day 1 of each course (if IT methotrexate is not administered).

Patients are followed every 2 months for 2 years, every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 260 patients will be accrued for this study within 3.1 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of B-cell precursor acute lymphoblastic leukemia

  * Registered on POG-9900 Classification Study
* Registered within 7 days of documenting complete response after induction on day 29 or, if 2 more weeks of induction are required, no later than day 49
* Classified as high risk:

  * No simultaneous trisomy 4 and 10
  * No TEL-AML1 gene
  * Meets criteria for 1 of the following:

    * Any age with WBC > 100,000/mm^3

      * CNS and bone marrow evaluations required for those patients with WBC > 100,000/mm^3 who are within 24 months of initial diagnosis
    * Age over 12 (boys) or 16 (girls)
    * If younger, WBC must be 1 of the following:

      * Greater than 80,000/mm^3 (for boys age 8 or girls age 12)
      * Greater than 60,000/mm^3 (for boys age 9 or girls age 13)
      * Greater than 40,000/mm^3 (for boys age 10 or girls age 14)
      * Greater than 20,000/mm^3 (for boys age 11 or girls age 15)
  * At least one of the following:

    * CNS 3 disease (CSF WBC at least 5/microliter with blasts present)
    * Testicular leukemia
    * MLL gene rearrangements

PATIENT CHARACTERISTICS:

Age:

* 1 to 21

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* See Disease Characteristics

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 276 (Actual)
Dates: Start 2000-03; Primary Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Augmented Berlin Frankfurt Muenster (BFM) therapy is superior to ALinC 14/15 therapy
  To determine for patients at high risk for treatment failure if the augmented Berlin Frankfurt Muenster (BFM) therapy is superior to ALinC 14/15 therapy, on the basis of historical controls.

CONTACTS AND LOCATIONS:
Overall Officials: William P. Bowman, MD, Study Chair — Cook Children's Medical Center - Fort Worth
Locations (20):
- United States (20):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Albert Einstein Clinical Cancer Center, The Bronx, New York
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Doernbecher Children's Hospital, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington

REFERENCES:
- [Background] Chen IM, Harvey RC, Mullighan CG, Gastier-Foster J, Wharton W, Kang H, Borowitz MJ, Camitta BM, Carroll AJ, Devidas M, Pullen DJ, Payne-Turner D, Tasian SK, Reshmi S, Cottrell CE, Reaman GH, Bowman WP, Carroll WL, Loh ML, Winick NJ, Hunger SP, Willman CL. Outcome modeling with CRLF2, IKZF1, JAK, and minimal residual disease in pediatric acute lymphoblastic leukemia: a Children's Oncology Group study. Blood. 2012 Apr 12;119(15):3512-22. doi: 10.1182/blood-2011-11-394221. Epub 2012 Feb 24. PMID 22368272
- [Background] Rabin KR, Gramatges MM, Borowitz MJ, Palla SL, Shi X, Margolin JF, Zweidler-McKay PA. Absolute lymphocyte counts refine minimal residual disease-based risk stratification in childhood acute lymphoblastic leukemia. Pediatr Blood Cancer. 2012 Sep;59(3):468-74. doi: 10.1002/pbc.23395. Epub 2011 Nov 18. PMID 22102553
- [Background] Yang JJ, Cheng C, Yang W, Pei D, Cao X, Fan Y, Pounds SB, Neale G, Trevino LR, French D, Campana D, Downing JR, Evans WE, Pui CH, Devidas M, Bowman WP, Camitta BM, Willman CL, Davies SM, Borowitz MJ, Carroll WL, Hunger SP, Relling MV. Genome-wide interrogation of germline genetic variation associated with treatment response in childhood acute lymphoblastic leukemia. JAMA. 2009 Jan 28;301(4):393-403. doi: 10.1001/jama.2009.7. PMID 19176441
- [Background] Borowitz MJ, Devidas M, Hunger SP, et al.: Prognostic signficance of end consolidation minimal residual disease (MRD) in childhood acute lymphoblastic leukemia (ALL): A report from the Children's Oncology Group (COG). [Abstract] J Clin Oncol 26 (Suppl 15): A-10000, 2008.
- [Background] Borowitz MJ, Devidas M, Hunger SP, Bowman WP, Carroll AJ, Carroll WL, Linda S, Martin PL, Pullen DJ, Viswanatha D, Willman CL, Winick N, Camitta BM; Children's Oncology Group. Clinical significance of minimal residual disease in childhood acute lymphoblastic leukemia and its relationship to other prognostic factors: a Children's Oncology Group study. Blood. 2008 Jun 15;111(12):5477-85. doi: 10.1182/blood-2008-01-132837. Epub 2008 Apr 3. PMID 18388178
- [Background] Davies SM, Borowitz MJ, Rosner GL, Ritz K, Devidas M, Winick N, Martin PL, Bowman P, Elliott J, Willman C, Das S, Cook EH, Relling MV. Pharmacogenetics of minimal residual disease response in children with B-precursor acute lymphoblastic leukemia: a report from the Children's Oncology Group. Blood. 2008 Mar 15;111(6):2984-90. doi: 10.1182/blood-2007-09-114082. Epub 2008 Jan 8. PMID 18182569
- [Background] Harvey RC, Mullighan CG, Wang X, Dobbin KK, Davidson GS, Bedrick EJ, Chen IM, Atlas SR, Kang H, Ar K, Wilson CS, Wharton W, Murphy M, Devidas M, Carroll AJ, Borowitz MJ, Bowman WP, Downing JR, Relling M, Yang J, Bhojwani D, Carroll WL, Camitta B, Reaman GH, Smith M, Hunger SP, Willman CL. Identification of novel cluster groups in pediatric high-risk B-precursor acute lymphoblastic leukemia with gene expression profiling: correlation with genome-wide DNA copy number alterations, clinical characteristics, and outcome. Blood. 2010 Dec 2;116(23):4874-84. doi: 10.1182/blood-2009-08-239681. Epub 2010 Aug 10. PMID 20699438
- [Background] Yang JJ, Yang W, Cheng C, et al.: Genetically defined racial differences underlie risk of relapse in childhood acute lymphoblastic leukemia. [Abstract] Blood 112 (11): A-14, 2008.
- [Result] Bowman WP, Larsen EL, Devidas M, Linda SB, Blach L, Carroll AJ, Carroll WL, Pullen DJ, Shuster J, Willman CL, Winick N, Camitta BM, Hunger SP, Borowitz MJ. Augmented therapy improves outcome for pediatric high risk acute lymphocytic leukemia: results of Children's Oncology Group trial P9906. Pediatr Blood Cancer. 2011 Oct;57(4):569-77. doi: 10.1002/pbc.22944. Epub 2011 Feb 25. PMID 21360654
- [Result] Zhang J, Mullighan CG, Harvey RC, Wu G, Chen X, Edmonson M, Buetow KH, Carroll WL, Chen IM, Devidas M, Gerhard DS, Loh ML, Reaman GH, Relling MV, Camitta BM, Bowman WP, Smith MA, Willman CL, Downing JR, Hunger SP. Key pathways are frequently mutated in high-risk childhood acute lymphoblastic leukemia: a report from the Children's Oncology Group. Blood. 2011 Sep 15;118(11):3080-7. doi: 10.1182/blood-2011-03-341412. Epub 2011 Jun 16. PMID 21680795
- [Result] Harvey RC, Mullighan CG, Chen IM, Wharton W, Mikhail FM, Carroll AJ, Kang H, Liu W, Dobbin KK, Smith MA, Carroll WL, Devidas M, Bowman WP, Camitta BM, Reaman GH, Hunger SP, Downing JR, Willman CL. Rearrangement of CRLF2 is associated with mutation of JAK kinases, alteration of IKZF1, Hispanic/Latino ethnicity, and a poor outcome in pediatric B-progenitor acute lymphoblastic leukemia. Blood. 2010 Jul 1;115(26):5312-21. doi: 10.1182/blood-2009-09-245944. Epub 2010 Feb 4. PMID 20139093
- [Result] Kang H, Chen IM, Wilson CS, Bedrick EJ, Harvey RC, Atlas SR, Devidas M, Mullighan CG, Wang X, Murphy M, Ar K, Wharton W, Borowitz MJ, Bowman WP, Bhojwani D, Carroll WL, Camitta BM, Reaman GH, Smith MA, Downing JR, Hunger SP, Willman CL. Gene expression classifiers for relapse-free survival and minimal residual disease improve risk classification and outcome prediction in pediatric B-precursor acute lymphoblastic leukemia. Blood. 2010 Feb 18;115(7):1394-405. doi: 10.1182/blood-2009-05-218560. Epub 2009 Oct 30. PMID 19880498
- [Result] Mullighan CG, Morin R, Zhang J, et al.: Next generation transcriptomic resequencing identifies novel genetic alterations in high-risk (HR) childhood acute lymphoblastic leukemia (ALL): A report from the Children's Oncology Group (COG) HR ALL TARGET Project. [Abstract] Blood 114 (22): A-704, 2009.
- [Result] Zhang J, Mullighan CG, Harvey RC, et al.: Mutations in the RAS signaling, B-cell development, TP53/RB1, and JAK signaling pathways are common in high risk B-precursor childhood acute lymphoblastic leukemia (ALL): A report from the Children's Oncology Group (COG) High-Risk (HR) ALL TARGET Project. [Abstract] Blood 114 (22): A-85, 2009.
- [Result] Harvey RC, Davidson GS, Wang X, et al.: Expression profiling identifies novel genetic subgroups with distinct clinical features and outcome in high-risk pediatric precursor B acute lymphoblastic leukemia (B-ALL). A Children's Oncology Group study. [Abstract] Blood 110 (11): A-1430, 2007.
- [Result] Kang H, Bedrick EJ, Chen IM, et al.: Molecular classifiers for prediction of minimal residual disease (MRD) and event free survival (EFS) improve risk assignment at diagnosis in pediatric high-risk B precursor acute lymphoblastic leukemia (ALL): a Childrens Oncology Group study. [Abstract] Blood 110 (11): A-1422, 2007.
- [Result] Borowitz MJ, Devidas M, Bowman WP, et al.: Prognostic significance of minimal residual disease (MRD) in children with high risk acute lymphoblastic leukemia(ALL): a Children's Oncology Group study. [Abstract] Blood 106 (11): A-85, 2005.
- [Derived] Fernandez CA, Smith C, Yang W, Date M, Bashford D, Larsen E, Bowman WP, Liu C, Ramsey LB, Chang T, Turner V, Loh ML, Raetz EA, Winick NJ, Hunger SP, Carroll WL, Onengut-Gumuscu S, Chen WM, Concannon P, Rich SS, Scheet P, Jeha S, Pui CH, Evans WE, Devidas M, Relling MV. HLA-DRB1*07:01 is associated with a higher risk of asparaginase allergies. Blood. 2014 Aug 21;124(8):1266-76. doi: 10.1182/blood-2014-03-563742. Epub 2014 Jun 26. PMID 24970932
- [Derived] Yang JJ, Cheng C, Devidas M, Cao X, Campana D, Yang W, Fan Y, Neale G, Cox N, Scheet P, Borowitz MJ, Winick NJ, Martin PL, Bowman WP, Camitta B, Reaman GH, Carroll WL, Willman CL, Hunger SP, Evans WE, Pui CH, Loh M, Relling MV. Genome-wide association study identifies germline polymorphisms associated with relapse of childhood acute lymphoblastic leukemia. Blood. 2012 Nov 15;120(20):4197-204. doi: 10.1182/blood-2012-07-440107. Epub 2012 Sep 24. PMID 23007406